CLINICAL TRIAL: NCT07322640
Title: Play Therapy With Gamified Biofeedback in Children With Autism Spectrum Disorder: A Randomized Clinical Trial
Brief Title: Play Therapy With Gamified Biofeedback in Children With Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luiz Alexandre Viana Magno (Other)
Responsible Party: Sponsor-Investigator, Luiz Alexandre Viana Magno, Principal Investigator, Faculdade de Ciências Médicas de Minas Gerais
Organization: Faculdade de Ciências Médicas de Minas Gerais (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 92066625.6.0000.5134
Record Dates: First submitted 2025-12-05; First posted 2026-01-07 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Autism Spectrum Disorder
Keywords: autism spectrum disorder; play therapy; biofeedback; emotional regulation; heart rate variability; Wearable Electronic Devices; children
MeSH Terms: conditions — Autism Spectrum Disorder; Emotional Regulation | interventions — Play Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Play Therapy + Gamified Biofeedback (Experimental): Children receive 8 weekly 50-minute individual sessions consisting of 35 minutes of child-centered play therapy followed by 15 minutes of gamified biofeedback using a heart-rate armband that adjusts game difficulty in real time plus continuous physiological monitoring with a wristband (HRV, EDA, skin temperature, accelerometry, respiratory rate). The biofeedback games become easier when the child successfully uses calming strategies.
  Interventions: Behavioral: Gamified Biofeedback; Behavioral: Play Therapy
- Play Therapy Alone (Active Comparator): Children receive 8 weekly 50-minute individual sessions identical in structure and duration to the experimental arm (35 minutes of child-centered play therapy). During the final 15 minutes they play the same tablet-based games as the experimental group, but with the biofeedback function deactivated and wearing the devices only for equivalence of contact; no real-time physiological feedback is provided.
  Interventions: Behavioral: Play Therapy; Behavioral: Deactivated Biofeedback

INTERVENTIONS:
Behavioral: Gamified Biofeedback — Participants receive 8 weekly 15-minute of gamified biofeedback using a non-invasive heart-rate monitor armband connected to a tablet-based platform. The games increase in difficulty when heart rate rises (indicating emotional arousal) and become easier when the child successfully applies calming strategies such as slow breathing or brief pauses. A second wearable wristband continuously records heart-rate variability, electrodermal activity, peripheral skin temperature, accelerometry, and respiratory rate for objective physiological monitoring throughout the biofeedback segment.
  Arms: Play Therapy + Gamified Biofeedback
Behavioral: Play Therapy — Participants receive 8 weekly 50-minute individual sessions with therapist of a play-based approach aimed at promoting joint attention, shared engagement, symbolic play, and emotional self-regulation. Toys will be selected according to the child's individual interests and tailored to their level of play development, incorporating both already mastered skills and emerging skills. Within these routines, strategies will be implemented such as: intentional pauses to encourage communicative initiation; expansion of play narratives to increase complexity and flexibility; balanced turn-taking to reinforce social reciprocity; modeling and positive reinforcement of gestures and verbal/nonverbal communication; and integration of emotional regulation techniques within the play context, facilitating the generalization of these skills to other environments.
Behavioral: Deactivated Biofeedback — Children will engage in the interactive play-based games used in the active biofeedback condition. The biofeedback device will be installed and worn. However, the biofeedback functionality will be deactivated and no physiological feedback will be provided to or influence the child during gameplay.
  Arms: Play Therapy Alone

SUMMARY:
This clinical trial tests whether combining regular play therapy with gamified biofeedback helps children with autism spectrum disorder better regulate their emotions and improve social skills, compared to play therapy alone. Sixty-eight children will be randomly assigned to 8 weekly 50-minute sessions: one group receives play therapy only, while the other receives play therapy plus real-time biofeedback using a comfortable armband that turns heart-rate calming into fun game rewards. Parents and teachers will complete short questionnaires before and after the study. All activities are playful, safe, and designed to feel natural and enjoyable for children with autism.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a neurodevelopmental condition characterized by persistent difficulties in social communication and interaction, restricted interests, and repetitive behaviors. Even in children with ASD level 1 (requiring support) who have normal or high cognitive abilities, emotional dysregulation is one of the most significant and persistent challenges. These children frequently experience intense physiological arousal in response to everyday sensory or social stimuli, yet they struggle to recognize, interpret, and self-regulate their emotional states. Traditional behavioral and developmental therapies improve communication and reduce repetitive behaviors, but emotional dysregulation often remains a major barrier to social participation, learning, and family well-being, contributing to frequent anxiety, and long-term mental health risks.

This single-center, pragmatic, parallel-group, single-blind (outcome assessor) randomized clinical trial aims to determine whether integrating real-time gamified biofeedback with standard child-centered play therapy produces greater improvements in emotional regulation and socioemotional skills than play therapy alone in children aged 6-10 years diagnosed with ASD level 1 according to DSM-5 criteria.

A total of 68 children will be consecutively recruited from the outpatient clinic of the Faculdade de Ciências Médicas de Minas Gerais (FCMMG), Belo Horizonte, Brazil. After obtaining written informed consent from parents/legal guardians and child assent, participants will be randomly allocated in a 1:1 ratio (using computer-generated randomization) to one of two interventions delivered over 12 weeks in weekly 50-minute individual sessions conducted by the same psychologist experienced in autism spectrum disorder.

Both groups receive identical child-centered play therapy focused on fostering joint attention, symbolic play, reciprocal interaction, and emotional co-regulation in a sensory-friendly room adapted for children with autism. The experimental group additionally receives gamified biofeedback (heart-rate monitor armband that adjusts game difficulty based on arousal level, rewarding successful calming strategies) and continuous physiological monitoring with the a FDA-cleared research device recording heart-rate variability, electrodermal activity, peripheral skin temperature, accelerometry, and respiratory rate). The control group plays the same tablet games but with the biofeedback function deactivated (sham condition).

Blinded assessments are conducted at baseline and immediately after the intervention. The primary outcome is the change in emotion regulation scores. Secondary outcomes include changes in sociability, behavior, parenting stress, and exploratory correlations between physiological biomarkers and clinical improvements. The study follows CONSORT guidelines and has been approved by the institutional ethics committee (CEP-FCMMG).

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 years and 10 years
* Formal diagnosis of autism spectrum disorder (ASD) level 1 according to DSM-5 criteria, documented by a qualified professional
* Signed informed consent by parent/legal guardian and child assent

Exclusion Criteria:

* Severe psychiatric comorbidities (e.g., psychosis, severe obsessive-compulsive disorder)
* Uncontrolled epilepsy or contraindication to biofeedback procedures
* Severe intellectual disability that prevents interaction with tablet-based games or biofeedback
* Severe or decompensated systemic medical conditions (e.g., active cancer, uncontrolled cardiac disease, uncontrolled diabetes)
* Change in dose or initiation of any psychotropic medication within 4 weeks prior to enrollment

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Emotion Regulation Checklist (ERC) total score | Baseline and 8 weeks of intervention
  Parent-rated emotional regulation measured by the Brazilian version of the Emotion Regulation Checklist (ERC). The ERC comprises the scales of Emotion Regulation (Range 8 to 32) andf Emotional Lability/Negativity (Range 15 to 60). An adaptive emotion regulation total score (range 23 to 92) is presented where a higher score is indicative of good emotion regulation and lower scores indicative of poor emotion regulation. This score is calculated by the sum of the emotion regulation scale and the inverse of the emotional lability/negativity scale.

SECONDARY OUTCOMES:
Change in Social Responsiveness Scale (SRS-2) (parent form) | Baseline and 8 weeks of intervention
  Parent-reported Brazilian version of the Social Responsiveness Scale, Second Edition (SRS-2), Parent Form, which assesses the severity of social impairment associated with autism spectrum symptoms. All items are rated on a 4-point Likert scale anchored by not true and almost always true, where high scores indicate greater dysfunction. Raw scores are converted into T-scores for interpretation.
Change in Social Responsiveness Scale (SRS-2) (teacher form) | Baseline and 8 weeks of intervention
  Teacher-reported scores in the Social Responsiveness Scale, Second Edition (SRS-2), Teacher Form, which measures social functioning in the school context. All items are rated on a 4-point Likert scale anchored by not true and almost always true, where high scores indicate greater dysfunction. Raw scores are converted into T-scores for interpretation.
Change in Child Behavior Checklist (CBCL 6/18) | Baseline and 8 weeks of intervention
  Parent-reported Brazilian version of Child Behavior Checklist (CBCL 6/18) is a caregiver-reported measure designed to assess behavioural and emotional problems in children and young people aged 6-18 years. The study will measure the problem behaviour scale, wich contains eight subscales that can be grouped into two higher-order factors, known as the internalising and externalising behaviours. By summing up all the problem items, a Total Problems score can also be computed. Higher scores indicate greater problems.
Change in Parenting Stress Index (PSI-4 SF) | Baseline and 8 weeks of intervention
  The Parenting Stress Index-Fourth Edition, Short Form (PSI-4 SF) assesses overall parenting stress. The total score ranges from 36 to 180, with higher scores indicating greater parenting stress (worse outcome).

OTHER OUTCOMES:
Correlation between physiological parameters and changes in clinical scales | Session-by-session physiological patterns across the intervention period (Baseline through Week 8)
  hysiological data will be collected during each intervention session, including heart rate variability (HRV), electrodermal activity (EDA), and skin temperature. These measures will be used to characterize session-by-session patterns and within-week changes in autonomic regulation from baseline through the end of the 8-week intervention period. Outcomes will reflect temporal trends and variability in physiological responses across sessions rather than a single summary score.

CONTACTS AND LOCATIONS:
Locations (1):
- Ambulatório da Faculdade de Ciências Médicas de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including data dictionaries) that underlie the results reported in the primary publication (including the primary and secondary outcome measures, baseline characteristics, and adverse events) will be made available upon reasonable request beginning 6 months and ending 5 years following article publication. Data will be shared with researchers who provide a methodologically sound proposal and have appropriate ethical approval. Requests should be directed to the Principal Investigator.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 6 months after publication - 5 years after publication
Access Criteria: Researchers must submit a brief research proposal and sign a data access agreement. Data will be shared via secure file transfer after approval by the Principal Investigator.